CLINICAL TRIAL: NCT03116958
Title: MyOSA : Management and Treatment of Patients With Obstructive Sleep Apnea Syndrome(OSAS) Through a Telemedicine System
Acronym: MyOSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: Fundació Eurecat (Other)
Responsible Party: Principal Investigator, Ferran Barbe, Head of Respiratory department at Hospital Universitari Arnau de Vilanova, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SEPAR 2016
Record Dates: First submitted 2017-04-03; First posted 2017-04-17 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Sleep Apnea Syndrome
Keywords: CPAP compliance; Telemedicine integrated platform; Standard management; Cost-effectiveness
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (Active Comparator): Patients diagnosed as OSA, treated with CPAP and followed up in sleep unit as per usual care.
  Patients will be fitted with a mask and given a CPAP and instructed on how to use the device. Each CPAP machine will be provided with a modem sending daily compliance and adherence information to MyOSA web site but no intervention based on these data is planned in this group. All patients will be visited at 1,3 and 6 months at sleep unit. Patients will be checked about progress and adherence to therapy and any problems with their machine. Information will be downloaded from their machines (CPAP adherence, applied CPAP pressure, mask leak, and residual respiratory events…).
  Interventions: Device: CPAP + Standard care
- Telemedicine (Experimental): Patients diagnosed as OSA and treated with CPAP, followed up in sleep unit, adding a telemedicine integrated system.
  Patients will be fitted with a mask , given a CPAP, and instructed on how to use the device. Using patients' baseline and initial follow-up data a software will provide a prediction of CPAP compliance at 6 months, and propose personalized interventions to increase compliance (smartphone app). All patients will be visited at 3 and 6 months at sleep unit. Patients will be checked about progress and adherence to therapy and any problems with their machine.
  Interventions: Device: CPAP + Telemedicine

INTERVENTIONS:
Device: CPAP + Standard care — CPAP device + Standard management at Sleep Unit. According to Spanish Respiratory Society guidelines during 6 months
  Arms: Standard care
Device: CPAP + Telemedicine — CPAP+ telemedicine approach. Patients followed up at Sleep Unit according to Spanish Respiratory Society guidelines during 6 months.
  Arms: Telemedicine

SUMMARY:
The purpose of this study is to improve CPAP treatment compliance of Obstructive Sleep Apnea Syndrome using an integrated telemedicine platform (MyOSA system)

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is defined by the presence of repetitive episodes of upper airways collapse during sleep, leading to nocturnal hypoxemia, sleep fragmentation and daytime sleepiness. When untreated, OSA is a risk factor for arterial hypertension , cardiovascular and cerebrovascular diseases, road accidents and a worse quality of life. The application of a continuous positive airways pressure (CPAP) represents the first line therapy in patients with moderate to severe OSA. CPAP treatment improves daytime sleepiness and oxygen saturation, reduces cardiovascular risk, ameliorates neurobehavioral performance, improves quality of life and reduces road accidents. Despite its demonstrated efficacy, CPAP effectiveness is significantly limited by poor adherence. A closer follow up could improve CPAP adherence but it would take up more work and additional costs for sleep units.

So, on that account, the investigators propose a study to evaluate the effect of adding a telemedicine approach to traditional follow up on CPAP treatment compliance, patients' satisfaction and follow-up costs.

Telemedicine will be provided by an integrated platform composed by a web site (https://www.myosa.net/menu/login.aspx) and a smartphone application.

Methods:

Design: Prospective randomised clinical study. Follow up: 6 months. Participants: 60 patients diagnosed as OSA at St. Maria's Hospital (Sleep Unit) and requiring CPAP treatment.

Randomization: Patients will be randomized into two groups differing in CPAP treatment management (standard care vs. telemedicine). Patients of both groups will be visited in Sleep Unit at 3st and 6th month after starting CPAP treatment. The CPAP machine of both groups will be provided with a modem sending daily information about CPAP treatment compliance and adherence to MyOSA web site (this kind of information will only be actively used during the follow-up in the telemedicine group).

Intervention:

Group 1- Telemedicine Patients will be fitted with a mask , given a CPAP, and instructed on how to use the device. An intelligent software specifically developed for this project will be integrated in the web site. Using patients' baseline data (sociodemographic characteristics, presence of comorbidities, quality of life, sleepiness, pharmacologic treatment, toxic habits), the software will be capable to provide an initial prediction of the expected CPAP compliance at 6 months. Then, the real data about patients' treatment compliance sent on daily base by the CPAP machine will train the software improving the level of confidence of the prediction. Based on the prediction of compliance at six months, the software will provide specific and personalized interventions to modify or maintain this prediction. Interventions will be administered to the patients through a smartphone application connected to the web site and specifically developed for this study (MyOSA-App). Using the mobile-app patients will receive information about their own CPAP compliance and advice on how to improve compliance. All patients will be visited at 3 and 6 months at sleep unit. Patients will be checked about progress and adherence to therapy and any problems with their machine.

Group 2- Standard care Patients will be fitted with a mask and given a CPAP and instructed on how to use the device. Each CPAP machine will be provided with a modem sending daily compliance and adherence information to MyOSA web site but no intervention based on these data is planned in this group. All patients will be visited at 1, 3 and 6 months at sleep unit. Patients will be checked about progress and adherence to therapy and any problems with their machine. Information will be downloaded from their machines (CPAP adherence, applied CPAP pressure, mask leak, and residual respiratory events…).

ELIGIBILITY:
Inclusion Criteria:

* Men and Women over 18 years old
* Diagnosed as OSA and requiring CPAP treatment
* Good knowledge of the use of a smartphone
* Written informed consent form signed

Exclusion Criteria:

* Patients with impaired lung function (overlap syndrome, obesity hypoventilation syndrome, and restrictive disorders)
* Severe heart failure
* Severe chronic pathology associated
* Psychiatric disorder
* Periodic leg movements
* Pregnancy
* Other dyssomnias or parasomnias
* Patients already treated with CPAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
CPAP compliance | 6 months
  Number of hours of use per day of CPAP according to the internal clock of the CPAP device

SECONDARY OUTCOMES:
CPAP adherence | 6 months
  Numbers of night with more than 4 hours of use
Patients' perceived ease of use of the telemedicine system | 6 months
  Patients in the telemedicine group will be asked to grade the perceived ease of use of the telemedicine platform using a questionnaire
Patients' perceived useful of the telemedicine system | 6 months
  Patients in the telemedicine group will be asked to grade the perceived useful of the telemedicine platform using a questionnaire
Patients' follow-up satisfaction | 6 months
  Patients of both group will be asked to grade their satisfaction with the follow up care provided by the sleep unit using a questionnaire.
Change from baseline in quality of life at 6 months | at baseline and 6 months
  EuroQOL health questionnaire will be used.
Change from baseline in daytime sleepiness at 6 months | at baseline and 6 months
  Epworth sleepiness scale will be used.
Abandons at 6 months | 6 months
  Number of patients lost at follow up at 6 months of CPAP therapy.
Cost effectiveness at 6 months | 6 months
  Costs in each group (telemedicine cost, CPAP carrying charge, number of visits and calls) will be compared.
Changes in treatment side effects | 6 months
Change in blood pressure at 6 months | at baseline and 6 months
Change in body mass index (in kg/m^2) at 6 months | at baseline and 6 months
Change from baseline in Visual analogue scale for quality of life at 6 months | at baseline and 6 months
  Visual analogue scale for quality of life will be used
Change in weight (in kg) at 6 months | at baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Barbe, MD, Principal Investigator — Hospital Arnau de Vilanova. IRB Lleida. CIBERes
Locations (1):
- Hospital Arnau de Vilanova, Lleida, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turino C, Benitez ID, Rafael-Palou X, Mayoral A, Lopera A, Pascual L, Vaca R, Cortijo A, Moncusi-Moix A, Dalmases M, Vargiu E, Blanco J, Barbe F, de Batlle J. Management and Treatment of Patients With Obstructive Sleep Apnea Using an Intelligent Monitoring System Based on Machine Learning Aiming to Improve Continuous Positive Airway Pressure Treatment Compliance: Randomized Controlled Trial. J Med Internet Res. 2021 Oct 18;23(10):e24072. doi: 10.2196/24072. PMID 34661550
- [Derived] Rafael-Palou X, Turino C, Steblin A, Sanchez-de-la-Torre M, Barbe F, Vargiu E. Comparative analysis of predictive methods for early assessment of compliance with continuous positive airway pressure therapy. BMC Med Inform Decis Mak. 2018 Sep 18;18(1):81. doi: 10.1186/s12911-018-0657-z. PMID 30227856